CLINICAL TRIAL: NCT06617130
Title: The Efficacy of Amino Acid Supplementation in Treating Environmental Enteric Dysfunction Among Children At Risk of Malnutrition
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kamuzu University of Health Sciences (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P.02/23/3992
Record Dates: First submitted 2024-09-16; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-06

CONDITIONS: Amino Acid, Stunting, Environmental Enteric Dysfunction
MeSH Terms: conditions — Growth Disorders | interventions — Amino Acids, Essential

STUDY DESIGN:
Intervention Model Description: We hypothesize that adding 12 mg/day of indispensable amino acids (IAA) to corn-soy blend blended flour porridge will reduce gut permeability amongst 6-36 month old rural Malawian children at risk of stunting compared to providing only corn-soy blended flour porridge without addition of indispensable amino acids for a period of 4 weeks.
  This will be a randomized, controlled open label parallel group efficacy clinical trial. Eligible children will be identified through a Demographic Surveillance System implemented by the study group at Mangochi district hospital. 66 children meeting set criteria will be randomised to receive corn-soy blended flour porridge (control group) or corn-soy blended flour porridge to which is added indispensable amino acids. The standard complementary food will provide 30% daily energy requirement while the amino acids in the intervention group will provide 1.5 times the estimated average requirement (EAR) for a healthy child.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- corn soy bean flour porridge with added indespensable amino acids (Active Comparator): Children in the intervention arm will receive corn-soy blended flour porridge mixed with IAA. The CSB flour will be packed in 1kg packets while the IAA will be packed in small plastic bags. Parent/caretakers will be taught how to prepare complementary porridge and will be provided utensils to estimate amounts of porridge to give to the child. Pre-weighed IAA will be provided so that mothers can mix the IAA to the prepared CSB porridge.
  The amount of porridge to be given to the child is estimated at 75g cooked porridge or 5 tablespoons of porridge. Likuni porridge is estimated to provide 403kcal per 100g when prepared using a standard recipe (Malawi Food and Nutrient Database). Based on the age range of the participating children we aim to provide an average of 250-302 kcal per child per day.
  Interventions: Dietary Supplement: Corn soy bean blended flour porridge plus indispensable amino acid
- Corn soy bean flour porridge (Other): Children in the control arm children will receive corn-soy blended flour porridge only. The CSB flour will be packed in 1kg packets. Parent/caretakers will be taught how to prepare complementary porridge and will be provided utensils to estimate amounts of porridge to give to the child.
  The amount of porridge to be given to the child is estimated at 75g cooked porridge or 5 tablespoons of porridge. Likuni porridge is estimated to provide 403kcal per 100g when prepared using a standard recipe (Malawi Food and Nutrient Database). Based on the age range of the participating children we aim to provide an average of 250-302 kcal per child per day.
  Interventions: Dietary Supplement: Corn soy bean blended flour porridge plus indispensable amino acid

INTERVENTIONS:
Dietary Supplement: Corn soy bean blended flour porridge plus indispensable amino acid — Protocol treatment will start within two weeks of enrollment to the study. Following the baseline study assessments, each participant will receive corn-soy bean blended flour porridge supplemented with IAAs (histidine, isoleucine, leucine, lysine, methionine, phenylalanine, threonine, tryptophan, and valine) dosed at 12g/d and providing 1.5 times the estimated average requirement (EAR) for a healthy child (Intervention group). The porridge will provide 30% daily energy requirement. The study foods will be taken once daily by the child with at least three observed feeding sessions per week over the 4 weeks of the study to assess compliance.
  Children in the control arm will receive corn-soy blended flour porridge without added amino acids.

SUMMARY:
A randomised controlled open label clinical trial to determine whether addition of indispensable amino acids (IAA) to standard complementary food will reduce occurrence of Environmental Enteric Dysfunction (EED) compared with provision of standard complementary food without IAA in healthy Malawian children aged 18-36 months with or without stunting.

ELIGIBILITY:
Inclusion Criteria:

* All children identified from the Mangochi DSS whose guardian/parent desires screening will be eligible for screening. This will first include age, weight, length, and MUAC assessment. If a participant meets age and anthropometric criteria, they will be invited to undergo full inclusion/exclusion criteria assessment, consent, and randomization.

In order to be eligible to participate in the study, an individual must meet all of the following criteria:

1. 18-36 months old (now agreed to by all countries)
2. Stunted (LAZ<-2)
3. Of either sex
4. Able and willing to undergo HIV testing
5. Parent, carer, or guardian able and willing to give written, informed consent
6. A positive HIV test result will not be an exclusion criterion.

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  1. Under 18 months of age
  2. Over 36 months old
  3. Wasted (weight-for-length Z-score less than -2)
  4. Overweight (weight-for-length Z-score greater than 2)
  5. Have had diarrhea (by self-report) in the preceding month
  6. Sibling or twin of another participating study child (2 children of different families in the same household are both eligible)
  7. Have any underlying condition other than HIV, which in the opinion of the investigator would put the subject at undue risk of failing study completion or would interfere with analysis of study results

Ages: 18 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
corn soy bean flour porridge with added indespensable amino acids | 30 days
  Primary Efficacy Endpoint:
  We hypothesize that adding 12mg IAA to corn-soy blended flour porridge provided to Malawian children aged 18-36 months with or without stunting will reduce gut permeability as measured by the Lactulose:Rhamonse ratio test when provided over 30 days compared to corn-soy blended flour porridge without added IAA.

SECONDARY OUTCOMES:
Corn soy bean flour porridge | 30 days
  We hypothesize that adding 12mg IAA to corn-soy blended flour porridge provided to Malawian children aged 18-36 months with or without stunting when provided over 30 days compared to corn-soy blended flour porridge without added IAA will:
  1. Increase gut digestive capacity
  2. Increase plasma protein absorption
  3. Reduce gut bacterial translocation
  4. Reduce gut bacterial damage
  5. Increase child weight
  6. Increase plasma circulating amino acids
  7. Increase gut microbial abundance and diversity
  8. Increase fat free mass index and fat free percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Kamuzu University of Health Sciences, Blantyre, Malawi

IPD SHARING:
Plan to Share IPD: Undecided
The Principal Investigator will determine authorship on primary and secondary publications of data derived from this trial and published by the PI's research group. De-identified data will be shared with PI approval beginning 6 months after primary trial publication with researchers that provide reasonable statistical analysis plans.